CLINICAL TRIAL: NCT02842255
Title: Calibration of a New Reflectance Oximeter.
Acronym: PATCHSANTESpO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 38RC15.098
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Volunteer
Keywords: Sleep apnea; Oximeter; Calibration; Oxygen partial pressure
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy volunteers (Experimental)
  Interventions: Device: Calibrate the oximeter ALTITRAINER200®

INTERVENTIONS:
Device: Calibrate the oximeter ALTITRAINER200® — During normoxic condition and four situations of hypoxia.

SUMMARY:
This study is about the development of a new medical device for the monitoring of of sleep disordered breathing. This device is developed by the CEA-LETI-LE2S and will be composed of an oximeter, an actimeter in order to measure the activity level of the subject, his state of sleeplessness/sleep, and a CO2 partial pressure transcutaneous sensor (PtcCO2).

Developing this device is realized in several steps : a study (ALMOST) is already in progress and its goal is to acquire a database of polysomnography to create automatic algorithms in order to detect respiratory disorders with this device under development.

The main goal of the study is to calibrate the oxymeter under development.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (both gender) aged between 18 to 50 years affiliated to a certain social security, that has given their free consent to participate to the study
* Subjets without any pathology known and not under medical treatment likely to suffer from controlled hypoxia at levels demanded in the protocol.
* Subjets having a regular practice of sport

Exclusion Criteria:

* Subjet non affiliated to a certain social security
* Smoker or person exposed to passive smoking
* History of acute mountain sickness or known sensitivity to hypoxia
* Any chronic pathology known, in particular pathologies behind high rates of methaemoglobin
* Pregnant, parturient or breastfeeding women, person deprived of liberty by judicial or administrative decision, person under a legally protected order and could'nt be included in clinical trials (persons mentioned in L1121-5 to L1121-8 of CSP).
* Subjets likely to not be cooperative or respectful of the inherent constraints to study participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Calibration of the oximeter in normoxic situation | 2 hours
  Measures with ALTITRAINER200® system Ambiant air : 98-96 % partial pressure in O2
Calibration of the oximeter in hypoxia situation | 2 hours
  Measures with ALTITRAINER200® system Situation 1 : 90 % (92-88%) partial pressure in O2 Situation 2 : 85% (87-83%) partial pressure in O2 Situation 3 : 80% (82-78%) partial pressure in O2 Situation 4 : 75%(77%-73%) partial pressure in O2

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Wuyam, Doctor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Berry RB, Budhiraja R, Gottlieb DJ, Gozal D, Iber C, Kapur VK, Marcus CL, Mehra R, Parthasarathy S, Quan SF, Redline S, Strohl KP, Davidson Ward SL, Tangredi MM; American Academy of Sleep Medicine. Rules for scoring respiratory events in sleep: update of the 2007 AASM Manual for the Scoring of Sleep and Associated Events. Deliberations of the Sleep Apnea Definitions Task Force of the American Academy of Sleep Medicine. J Clin Sleep Med. 2012 Oct 15;8(5):597-619. doi: 10.5664/jcsm.2172. PMID 23066376
- [Background] Dempsey JA, Veasey SC, Morgan BJ, O'Donnell CP. Pathophysiology of sleep apnea. Physiol Rev. 2010 Jan;90(1):47-112. doi: 10.1152/physrev.00043.2008. PMID 20086074
- [Background] Chouri-Pontarollo N, Borel JC, Tamisier R, Wuyam B, Levy P, Pepin JL. Impaired objective daytime vigilance in obesity-hypoventilation syndrome: impact of noninvasive ventilation. Chest. 2007 Jan;131(1):148-55. doi: 10.1378/chest.06-1159. PMID 17218569
- [Background] Becker HF, Piper AJ, Flynn WE, McNamara SG, Grunstein RR, Peter JH, Sullivan CE. Breathing during sleep in patients with nocturnal desaturation. Am J Respir Crit Care Med. 1999 Jan;159(1):112-8. doi: 10.1164/ajrccm.159.1.9803037. PMID 9872827
- [Background] Peppard PE, Young T, Palta M, Skatrud J. Prospective study of the association between sleep-disordered breathing and hypertension. N Engl J Med. 2000 May 11;342(19):1378-84. doi: 10.1056/NEJM200005113421901. PMID 10805822
- [Background] Perrin C, Unterborn JN, Ambrosio CD, Hill NS. Pulmonary complications of chronic neuromuscular diseases and their management. Muscle Nerve. 2004 Jan;29(1):5-27. doi: 10.1002/mus.10487. PMID 14694494
- [Background] Flemons WW, Reimer MA. Development of a disease-specific health-related quality of life questionnaire for sleep apnea. Am J Respir Crit Care Med. 1998 Aug;158(2):494-503. doi: 10.1164/ajrccm.158.2.9712036. PMID 9700127
- [Background] Nitzan M, Romem A, Koppel R. Pulse oximetry: fundamentals and technology update. Med Devices (Auckl). 2014 Jul 8;7:231-9. doi: 10.2147/MDER.S47319. eCollection 2014. PMID 25031547
- [Background] Mollard P, Bourdillon N, Letournel M, Herman H, Gibert S, Pichon A, Woorons X, Richalet JP. Validity of arterialized earlobe blood gases at rest and exercise in normoxia and hypoxia. Respir Physiol Neurobiol. 2010 Jul 31;172(3):179-83. doi: 10.1016/j.resp.2010.05.017. Epub 2010 May 21. PMID 20493971
- [Background] Richalet JP, Larmignat P, Poitrine E, Letournel M, Canoui-Poitrine F. Physiological risk factors for severe high-altitude illness: a prospective cohort study. Am J Respir Crit Care Med. 2012 Jan 15;185(2):192-8. doi: 10.1164/rccm.201108-1396OC. Epub 2011 Oct 27. PMID 22071330
- [Background] Savourey G, Launay JC, Besnard Y, Guinet-Lebreton A, Alonso A, Sauvet F, Bourrilhon C. Normo or hypobaric hypoxic tests: propositions for the determination of the individual susceptibility to altitude illnesses. Eur J Appl Physiol. 2007 May;100(2):193-205. doi: 10.1007/s00421-007-0417-8. Epub 2007 Feb 24. PMID 17323073
- [Background] Aguilaniu B, Maitre J, Diab S, Perrault H, Peronnet F. Detection of disturbances in pulmonary gas exchanges during exercise from arterialized earlobe PO2. Respir Physiol Neurobiol. 2011 Jun 30;177(1):30-5. doi: 10.1016/j.resp.2011.03.005. Epub 2011 Mar 17. PMID 21397053